CLINICAL TRIAL: NCT01155869
Title: Pilot Study of Depot Naltrexone in Alcohol-Dependent, Homeless Veterans
Brief Title: Pilot Study of Depot NTX in Homeless Veterans
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PPO 10-079
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-06

CONDITIONS: Alcohol Dependence
Keywords: alcohol dependence; homelessness; naltrexone
MeSH Terms: conditions — Alcoholism | interventions — vivitrol; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- XR-NTX (Experimental): Depot naltrexone (Vivitrol) 380 mg. IM monthly
  Interventions: Drug: Depot naltrexone
- Oral Naltrexone (Active Comparator): Naltrexone 50 mg tablet PO daily
  Interventions: Drug: Oral Naltrexone

INTERVENTIONS:
Drug: Depot naltrexone — Depot naltrexone 380 mg. IM monthly
  Other Names: Vivitrol
  Arms: XR-NTX
Drug: Oral Naltrexone — Naltrexone 50 mg tablet PO daily
  Other Names: Revia
  Arms: Oral Naltrexone

SUMMARY:
Almost 200,000 veterans are homeless each night, about one-quarter to one-third of homeless adults in the U.S. Half need treatment for a substance use disorder, usually alcohol dependence, but sobriety is often required to access alcohol treatment and housing services. A monthly injection of depot naltrexone is efficacious in reducing alcohol use, but it is expensive and restricted in many VA Medical Centers. Oral naltrexone is more available but seldom used because of adherence problems that limit effectiveness. This open-label pilot study would compare the effect of depot versus oral naltrexone to help twenty homeless, alcohol-dependent veterans decrease their drinking, achieve sobriety and qualify for housing services. This study's findings could expand access to effective medication-assisted alcohol treatment in the VA, and thus help homeless veterans with alcohol problems improve their drinking, housing status, and appropriate use of health services.

DETAILED DESCRIPTION:
Anticipated Impacts on Veteran's Healthcare. Ending homelessness among veterans is a major priority for VA. Veterans represent between one in four and one in three homeless adults. Almost 200,000 veterans are homeless each night. Rhode Island has the second highest per capita concentration of homeless persons in the United States and an estimated 2,000 homeless veterans. Half report unmet service needs related to substance use disorders. The VA is a major service provider to homeless persons and has developed innovative housing assistance programs. However, sobriety is required to access many housing services. Effective medication-assisted treatment for the alcohol-dependent, homeless population could improve their substance use, health care utilization and housing stability. If depot naltrexone is a useful tool for engaging alcohol-dependent, homeless veterans in effective treatment, a definitive study showing its effect would lead to fewer restrictions on depot naltrexone on the VA formulary, and expand access to effective medication-assisted treatment.

Project Background/Rationale. A dearth of residential long-term rehabilitation beds makes an initial period of sobriety necessary in order for homeless persons to access needed transitional sheltering in order to participate in outpatient alcohol treatment. Many alcohol-dependent homeless veterans find it difficult to achieve a period of sobriety. Clinical trials suggest that depot naltrexone is more efficacious than placebo in improving alcohol consumption among alcohol-dependent subjects, but depot naltrexone is expensive and has limited availability in many VA Medical Centers. Oral naltrexone is widely available but seldom used. This work seeks to examine the effect of depot versus oral naltrexone to help homeless alcohol dependent veterans.

Project Objectives. This open-label pilot study will compare the effect of 16-weeks of depot versus oral naltrexone among housing-seeking, alcohol dependent, homeless veterans. Outcomes will include alcohol consumption, housing stability, emergency department and hospital utilization, and substance abuse treatment participation. These preliminary data will evaluate the feasibility and effect size to allow the design of a larger, more definitive study of whether, compared to the oral naltrexone condition, the depot naltrexone group will experience: greater proportion of days abstinent and fewer drinks per drinking day; shorter time to achieve 30 days sobriety; more improvement in housing stability; fewer emergency department visits and hospitalizations and greater attendance at substance abuse treatment (number of visits attended).

Project Methods. Over 5 months, 20 homeless, alcohol dependent veterans will be recruited from the waiting lists for transitional or permanent housing at the Providence VA Medical Center. Using block randomization to stratify by current duration of abstinence (less than 7 days vs. 7 or more days) and sheltering (doubled-up/unsheltered/emergency vs. transitional sheltered), subjects will be assigned to either injection with depot naltrexone 380 mg. monthly or oral naltrexone 50 mg daily for 16 weeks. All will have medical visits with medication management counseling every 4 weeks with during the treatment period. Referrals will be made to needed services in keeping with standard practice. Research assessments at baseline and every 4 weeks through week 24 will assess alcohol consumption through self-report on calendar-based interviews, breathalyzer and liver enzyme testing. Primary outcomes will be alcohol consumption and time from randomization-to-30-day-sobriety. Secondary outcomes will include housing stability (across 5 ordered categories), emergency department and hospital utilization, and alcohol treatment participation from administrative data, CPRS abstracting and self-report.

ELIGIBILITY:
Inclusion Criteria:

1. Homeless per the federal definition (HEARTH Act, 2009), which includes individuals who lack a fixed, regular, and adequate nighttime residence; and those who have a primary nighttime residence that is a supervised publicly or privately operated shelter designed to provide temporary accommodations (including welfare hotels, congregate shelters, and transitional housing); an institution that provides a temporary residence for individuals intended to be institutionalized; and/or a public or private place not designed for, or ordinarily used as, a regular sleeping accommodation for human beings (including doubled up with a friend or family member).
2. Meet criteria for a DSM-IV diagnosis of alcohol abuse or dependence in the past year.
3. Last reported drink between 12 hours and 12 months prior, and BAC by breathalyzer of .08 or less.
4. Age between 18 and 64 years.
5. Eligible to receive VA services.
6. Willing to provide informed consent that will include all study procedures.
7. Those who report any opiate use in the past month must pass a naloxone challenge test (no sign of opiate withdrawal after IM injection of 0.8 mg naloxone).
8. If female of childbearing potential -- must be using adequate contraception.
9. Cognitively intact and showing no signs of delusional thought processes on the Short Blessed test (Callahan, 2002) and SCID checklist. Those with an untreated SMI and/or not capable of understanding the study due to an active cognitive impairment or delusional thought process will be excluded.
10. Speak English sufficiently to understand instructions and assessments.

Exclusion Criteria:

1. Untreated disorder that might make participation hazardous (e.g. untreated psychosis or bipolar disorder with mania on SCID checklist or significant suicide risk on Modified Scale of Suicidal Ideation (MSSI).
2. Use of contraindicated medications such as an opioid for a documented diagnosis or opiate maintenance.
3. Chronic pain condition or expected procedure during the study that is likely to require opioid analgesia.
4. Contraindicated medical conditions including pregnancy/lactation; liver failure or liver function test levels greater than three times normal; glaucoma; prior adverse reaction to naltrexone; life expectancy of less than 6 months or medical condition that will likely require skilled nursing facility care) within 6 months.
5. Stated plan to leave the area within 6 months of enrollment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Friedmann, MD MPH, Principal Investigator — VA Medical Center, Providence
Locations (1):
- VA Medical Center, Providence, Providence, Rhode Island, United States

REFERENCES:
- [Result] Friedmann PD, Mello D, Lonergan S, Bourgault C, O'Toole TP. Aversion to injection limits acceptability of extended-release naltrexone among homeless, alcohol-dependent patients. Subst Abus. 2013;34(2):94-6. doi: 10.1080/08897077.2012.763083. PMID 23577900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 215 potential subjects were approached over a 16-month period of recruitment; only 15 agreed to be screen after hearing of study procedures.
Pre-assignment Details: 5 were excluded (1 did not meet criteria for homelessness, 1 did not meet criteria for alcohol dependence, 1 had untreated delusional thinking, and 2 had opioid-requiring pain); 3 eligible participants did not appear for baseline interview and could not be found; only 7 were randomized.
Period: Overall Study
Arm/Group | XR-NTX | Oral Naltrexone
Started | 3 | 4
Completed | 0 | 3
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XR-NTX | Oral Naltrexone | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Weekly Self-reported Alcohol Consumption
Description: Mean number of standard drinks per week during the 24 week study. A standard drink is any drink that contains about 14 grams of pure alcohol, e.g. 12 ounces of beer, 5 ounces of wine or 1.5 ounces of spirits.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: standard drink
Arm/Group | XR-NTX | Oral Naltrexone
Number analyzed (Participants) | 3 | 4
standard drink | 0 (0) | 65 (10.6)

2. Secondary Outcome: Treatment Participation
Description: Percentage of total during-treatment study visits attended. This serves as a proxy for the number of months of treatment participation
Time Frame: 16 weeks
Measure: Number; unit: percentage of visits
Units Other Than Participants: Visits
Arm/Group | XR-NTX | Oral Naltrexone
Number analyzed (Participants) | 3 | 4
Number analyzed (Visits) | 12 | 16
percentage of visits | 33.3 | 87.5

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | XR-NTX | Oral Naltrexone
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XR-NTX (N=3) | Oral Naltrexone (N=4)
death (Investigations) | 1 (1) | 0 (0) — Pt missed appt for second injection and study interview. In trying to locate the subject, RA periodically checked CPRS. Record located in CPRS noted death.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XR-NTX (N=3) | Oral Naltrexone (N=4)
Arrest (Social circumstances) | 0 (0) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Emergency department visit

LIMITATIONS AND CAVEATS:
Only 15 of 215 alcohol-dependent, homeless veterans would consider a study that included an intramuscular injection of XR-NTX. Of 3 given XR-NTX, only 1 returned for injection #2. Aversion to injection likely contributed to poor acceptability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No